CLINICAL TRIAL: NCT02452697
Title: A Randomized Phase II Trial to Evaluate Progression-Free Survival Rates in Patients Receiving NK Cell-Enriched Donor Cell Infusions When Administered Alone or Administered With the TLR9 Agonist, DUK-CPG-001, From a 4-6/8 HLA-Matched Related or 7-8/8 HLA-Matched Donor Following Reduced Intensity or Non-Ablative Allogeneic Stem Cell Transplantation
Brief Title: Ph2 NK Cell Enriched DCIs w/wo RLR9 Agonist, DUK-CPG-001 From Donors Following Allogeneic SCT
Acronym: NK-DCI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cristina Gasparetto (Other)
Collaborators: Agilent Technologies, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Cristina Gasparetto, Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00057501; IND 16610 (Other: FDA)
Record Dates: First submitted 2015-02-06; First posted 2015-05-25 (Estimated); Results first posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-01

CONDITIONS: Myeloid Malignancies; Lymphoid Malignancies
Keywords: Nonmyeloablative; Stem Cell; Transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort A - NK cell enriched-DLI only (Active Comparator): Patients with a 7-8/8 human leukocyte antigen (HLA)-matched related or unrelated donor receiving natural killer (NK) cell enriched donor lymphocyte infusion (DLI) only
  Interventions: Biological: NK Cell enriched-DLI only
- Cohort A - NK-DLI + DUK-CPG-001 (Experimental): Patients with a 7-8/8 human leukocyte antigen (HLA)-matched related or unrelated donor receiving natural killer (NK) cell enriched donor lymphocyte infusion (DLI) and investigational DUK-CPG-001
  Interventions: Biological: NK-DLI + DUK-CPG-001
- Cohort B - NK cell enriched-DLI only (Active Comparator): Patients with a 4-6/8 human leukocyte antigen (HLA)-matched related donor receiving natural killer (NK) cell enriched donor lymphocyte infusion (DLI) only
  Interventions: Biological: NK Cell enriched-DLI only
- Cohort B - NK-DLI + DUK-CPG-001 (Experimental): Patients with a 4-6/8 human leukocyte antigen (HLA)-matched related donor receiving natural killer (NK) cell enriched donor lymphocyte infusion (DLI) and investigational DUK-CPG-001
  Interventions: Biological: NK-DLI + DUK-CPG-001

INTERVENTIONS:
Biological: NK Cell enriched-DLI only — The first NK cell-enriched DLI will be administered one to six months post transplant. The second NK cell-enriched DLI will be administered one to three months post the first infusion, in patients who have ≤ grade II aGVHD at the time of infusion and have not had unacceptable toxicities from the first infusion. Patients will continue on their stable dose of immunosuppressive agents started for therapy of acute GVHD before the NK cell-enriched DLI, and will not taper until at least 6 weeks following the each NK cell-enriched DLI (unless disease progression or patient toxicity from the agents requires earlier taper). The donor NK cells will be infused over 30 minutes intravenously.
  If signs of GVHD occur after NK cell-enriched DLI, immunosuppressive agents may be started.
  Arms: Cohort A - NK cell enriched-DLI only; Cohort B - NK cell enriched-DLI only
Biological: NK-DLI + DUK-CPG-001 — DUK-CPG-001 was synthesized by Agilent Technologies (Boulder, CO) in 2013. Bulk DUK-CPG-001 has been resuspended in normal saline with a final concentration of 10 mg/mL, aliquoted into 0.75 mL (7.5 mg) per tube and stored at -20oC in the Investigational Chemotherapy Service pharmacy at Duke. DUK-CPG-001 will be thawed at room temperature right before use and injected intravenously right after NK cell-enriched DLI. The drug will be used within 4 hours of thawing.
  On the day of NK cell-enriched DLI, for those patients who are randomized to receive DUK-CPG-001, 0.5 mL (5 mg) aliquots of DUK-CPG-001 will be dispensed to nurse. It will be thawed at room temperature right before use and injected intravenously right after NK cell-enriched DLI.
  Arms: Cohort A - NK-DLI + DUK-CPG-001; Cohort B - NK-DLI + DUK-CPG-001

SUMMARY:
This is a randomized, parallel phase II study to evaluate the rates of progression-free survival and unacceptable toxicity in patients receiving NK cell-enriched donor lymphocyte infusions (DLIs) when administered alone or administered with the TLR9 agonist, DUK-CPG-001, from a 7-8/8 HLA-matched related or unrelated donor (Cohort A) or 4-6/8 HLA-matched related donor (Cohort B) following reduced intensity or non-ablative allogeneic stem cell transplantation. Randomization will be stratified for disease types (myeloid versus lymphoid malignancies). Primary endpoints are analyzed separately in Cohort A and B.

Cohort A: 7-8/8 HLA-matched related or unrelated donor ("NK cell enriched-DLI only" arm or "NK cell enriched-DLI + DUK-CPG-001" arm)

Cohort B: 4-6/8 HLA-matched related donor ("NK cell enriched-DLI only" arm or "NK cell enriched-DLI + DUK-CPG-001" arm)

DETAILED DESCRIPTION:
This is a randomized, parallel phase II study to evaluate the rates of progression-free survival and unacceptable toxicity in patients receiving NK cell-enriched donor lymphocyte infusions (DLIs) when administered alone or administered with the TLR9 agonist, DUK-CPG-001, from a 7-8/8 HLA-matched related or unrelated donor (Cohort A) or 4-6/8 HLA-matched related donor (Cohort B) following reduced intensity or non-ablative allogeneic stem cell transplantation. Randomization will be stratified for disease types (myeloid versus lymphoid malignancies).

Patient prior to starting therapy Within 21 days prior to initiating therapy, patients will have an updated history and physical examination performed, lab tests, stool collection, and pregnancy test if the patient is a female of childbearing potential. Patients will have blood or marrow stored for analysis of immune function and chimerism. Tests documenting the patient's disease state are required at study entry as well (bone marrow aspirate/biopsy, blood studies, and/or radiographic tests such as CTs, MRI, PET scans as determined by treating physician,and as required for standardized response evaluations).

Donor apheresis and cell processing Donors will return to the center for a fresh collection of NK cells and they will not need growth factor mobilization. One collection will be used for each NK cell infusion. Cells will be transfused immediately after collection and processing or the next day. Cell processing will be performed in our cryopreservation lab according to SOP for collection, labeling and handling. The cells will be NK selected using a CD56 antibody (CliniMACS CD56 Reagent), CliniMACSplus instrument and CliniMACS tubing set provided by Miltenyi Biotec using the company protocol (Miltenyi Biotec Inc, Auburn, California). Pre and post processing cell count, viability, Hematopoietic Progenitor Cell Assay (HPCA) and flow analysis per SOP will be done.

Patient Evaluation Assessment of disease will use standardized criteria and shall include a careful examination of the studies needed to detect the disease (PET, radiographs, immuno phenotype, marrow, molecular studies etc). Restaging may be altered at the discretion of the transplant physician following the patient (who are all subinvestigators in this study) if the patient is felt to be progressing before these time points but the recommended restaging is q3 months for 1 year after the last NK-enriched DLI, q6 months for the next 2 years, then as indicated clinically. Immune reconstitution studies prior to and 1 and 7 days after each NK cell-enriched DLI, and 3, 6, and 12 months after the last NK-enriched DLI. Determination of chimerism (by short tandem repeat analysis in use in our DUKE HLA laboratory with a 2% sensitivity) just prior to each NK cell-enriched DLI, and 3, 6, 12 months after the last NK-enriched DLI.

Toxicity will be formally evaluated post infusion and a week later (more as determined by treatment team) and at a minimum of every other week through 6 weeks post infusion, then q3 months starting at 3 months post-second DLI for the first year. Assessments include history (specific to GI toxicity as well as overall new problems), physical exam, CBC, liver function tests (AST, ALT, bilirubin at a minimum), and Chemistry CS to include creatinine and BUN for toxicity assessment following the NCI common toxicity criteria (version 4) and standard GVHD criteria (appendix I). Further follow up will be required as needed if the patient has a toxicity due the transplant or infusion procedures. Patients with a grade 3 or greater toxicity due to the study will be seen every other week at a minimum until the toxicity is < grade 3, and then will be seen as clinically appropriate.

Stool Collection and Microbiome Analysis:

We will collect stool samples from patients at the following time points throughout the study: pre-DLI, day +7, pre-second DLI, day +7, then every 3 months post DLI for one year. Stool samples from patients may be stored at 4°C for up to 24 h before freezing at -80°C for batch analysis.

Patient NK cell infusion and CpG administration plan The target cell dose for NK cell-enriched DLI will be as many cells as can be collected with less than 0.5 x 106 CD3+ CD56- cells/kg patient weight in the 4-6/8 HLA-matched related setting and 1 x 106 CD3+ CD56- cells/kg patient weight in the 7-8/8 HLA-matched related or unrelated setting. The first NK cell-enriched DLI will be administered one to six months post transplant. The second NK cell-enriched DLI will be administered one to three months post the first infusion, in patients who have < grade II aGVHD at the time of infusion and have not had unacceptable toxicities that are at least possibly related to the previous DLI and resolved to grade 1 or less. The second DLI will NOT be administered in patient with ≥grade III aGVHD at the time of infusion or unacceptable toxicities at least possibly related to the first infusion. If patients have GVHD and were on immunosuppressive therapy at study entry, patients will continue on their stable dose of immunosuppressive agents started for therapy of acute GVHD before the NK cell-enriched DLI, and will not taper until at least 6 weeks following the each NK cell-enriched DLI (unless disease progression or patient toxicity from the agents requires earlier taper). The donor NK cells will be infused over 30 minutes. Diphenhydramine 25 mg iv or po, and Acetaminophen 650 mg po will be used prior to each reinfusion, unless there is a history of allergy or contraindication in the patient, in which case hydrocortisone 50mg IV will be used.

These cells are infused into the patient via a peripheral intravenous line or central line. If signs of GVHD occur after NK cell-enriched DLI, immunosuppressive agents (prednisone, cyclosporine, tacrolimus and/ or mycophenolate preferred first choices) may be started.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with hematologic diseases who have undergone T-cell depleted reduced intensity or non-ablative allogeneic transplantation, using a 7-8/8 HLA-matched related or unrelated donor or 4-6/8 HLA-matched related donor. This may include patients with a mixed chimeric state or disease persistence or at high risk of relapse.
2. Performance status must be ECOG PS 0, 1, or 2.
3. Donor cellular engraftment of at least 2.5% from the non-myeloablative procedure.
4. < Grade 2 acute GVHD at time of the first NK cell-enriched DLI. Patients with treated acute GVHD must be on a stable dose of therapy (no increase in immunosuppressive therapy for the 2 weeks before planned NK cell-enriched DLIs). The dosage/level of immunosuppressive therapy at the time of NK-DLIs should be no greater than 20 mg of prednisone daily or mycophenolate 500 mg bid daily or cyclosporine with a target level of 200 ng/mL or tacrolimus with a target level of 10 ng/mL.
5. Estimated survival of at least 8 weeks.
6. Age of >= 18 years.
7. Females of childbearing potential should have a negative serum beta-HCG test within 48 hours of beginning DLI and/or DUK-CPG-01 unless contraception is used after initial testing. A female of childbearing potential (FCBP) is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
8. Males must agree to use a medically acceptable form of birth control in order to be in this study and for 3 months after infusion

Exclusion Criteria:

1. Pregnant or lactating women.
2. Patients with other major medical or psychiatric illnesses, which the treating physician feels, could seriously compromise tolerance to this protocol.
3. Patients likely to have a significantly better durable response to allogeneic transplant alone (better than 60% progression free longer than 2 years) includes: those with myeloproliferative diseases or hemoglobinopathies with over 50% T cell subset engraftment (assessed around 100 days post transplant); It is not anticipated that any such patients would be transplanted within our program, however but those in first remission AML patients with good risk standard genetics or normal genetics with either NPM1 or CEBPA mutations, first chronic phase CML without kinase gene mutations, follicular lymphoma patients in first remission who only required 1 regimen to attain remission all would be excluded from this protocol.

HLA 4-6/8 matched related donor inclusion/exclusion criteria (criterion below are recommended but may evolve to follow current program standards) to be completed within 30 days of apheresis per standard guidelines

1. Adult donors must be an HLA 4-8/8 match with the patient and must be capable of providing informed consent.
2. Potential donors under the age of 18 must have a 'single patient exemption' approved by the IRB. The donor must provide assent and the donor's parent or guardian must provide permission for minor participation. Donors under the age of 18 who cannot assent based on their developmental stage will not be included.
3. Donor must not have any medical condition which would make apheresis more than a minimal risk, and should have the following:

   1. Family members will be considered for donation if they do not have a history of known cardiac problem and do not have abnormal cardiac findings by physical examination. Those with a history of cardiac problems or abnormal cardiac findings by physical examination should undergo a stress evaluation or be evaluated by a cardiologist and deemed eligible to donate.
   2. Documented bilirubin and hepatic transaminases of < 2.5 x ULN,
   3. Documented adequate hematologic parameters including a hematocrit > 35% for males and 33% for females, white blood cell count of >=3,000, and platelets >=80,000.
   4. FACT labs and final test results available prior to infusion into the patient. In the second donation from the donor, the FACT labs must be redrawn within 30 days of initiation of apheresis. Positive serologies are not repeated as they remain positive for lifetime.
4. Females of childbearing potential should have a negative serum beta-HCG test within 1 week of beginning apheresis. A female of childbearing potential (FCBP) is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months). A tubal ligation is adequate documentation that a patient is not of child bearing potential.

7-8/8 HLA matched unrelated donors will be matched at least as HLA -A, -B, C and -DRB1. Criterion for donation will be those allowing donation following the NMDP accepted donor criterion and program SOPs for the typical matched unrelated donors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-06-08 (Actual); Primary Completion 2022-07-23 (Actual); Study Completion 2024-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Gasparetto, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A - NK Cell Enriched-DLI Only: Patients with a 7-8/8 human leukocyte antigen (HLA)-matched related or unrelated donor receiving natural killer (NK) cell enriched donor lymphocyte infusion (DLI) only
  NK Cell enriched-DLI only: The first NK cell-enriched DLI will be administered one to six months post transplant. The second NK cell-enriched DLI will be administered one to three months post the first infusion, in patients who have ≤ grade II aGVHD at the time of infusion and have not had unacceptable toxicities from the first infusion. Patients will continue on their stable dose of immunosuppressive agents started for therapy of acute GVHD before the NK cell-enriched DLI, and will not taper until at least 6 weeks following the each NK cell-enriched DLI (unless disease progression or patient toxicity from the agents requires earlier taper). The donor NK cells will be infused over 30 minutes intravenously.
  If signs of GVHD occur after NK cell-enriched DLI, immunosuppressive agents may be started.
- Cohort A - NK-DLI + DUK-CPG-001: Patients with a 7-8/8 human leukocyte antigen (HLA)-matched related or unrelated donor receiving natural killer (NK) cell enriched donor lymphocyte infusion (DLI) and investigational DUK-CPG-001
  NK-DLI + DUK-CPG-001: DUK-CPG-001 was synthesized by Agilent Technologies (Boulder, CO) in 2013. Bulk DUK-CPG-001 has been resuspended in normal saline with a final concentration of 10 mg/mL, aliquoted into 0.75 mL (7.5 mg) per tube and stored at -20oC in the Investigational Chemotherapy Service pharmacy at Duke. DUK-CPG-001 will be thawed at room temperature right before use and injected intravenously right after NK cell-enriched DLI. The drug will be used within 4 hours of thawing.
  On the day of NK cell-enriched DLI, for those patients who are randomized to receive DUK-CPG-001, 0.5 mL (5 mg) aliquots of DUK-CPG-001 will be dispensed to nurse. It will be thawed at room temperature right before use and injected intravenously right after NK cell-enriched DLI.
- Cohort B - NK Cell Enriched-DLI Only: Patients with a 4-6/8 human leukocyte antigen (HLA)-matched related donor receiving natural killer (NK) cell enriched donor lymphocyte infusion (DLI) only
  NK Cell enriched-DLI only: The first NK cell-enriched DLI will be administered one to six months post transplant. The second NK cell-enriched DLI will be administered one to three months post the first infusion, in patients who have ≤ grade II aGVHD at the time of infusion and have not had unacceptable toxicities from the first infusion. Patients will continue on their stable dose of immunosuppressive agents started for therapy of acute GVHD before the NK cell-enriched DLI, and will not taper until at least 6 weeks following the each NK cell-enriched DLI (unless disease progression or patient toxicity from the agents requires earlier taper). The donor NK cells will be infused over 30 minutes intravenously.
  If signs of GVHD occur after NK cell-enriched DLI, immunosuppressive agents may be started.
- Cohort B - NK-DLI + DUK-CPG-001: Patients with a 4-6/8 human leukocyte antigen (HLA)-matched related donor receiving natural killer (NK) cell enriched donor lymphocyte infusion (DLI) and investigational DUK-CPG-001
  NK-DLI + DUK-CPG-001: DUK-CPG-001 was synthesized by Agilent Technologies (Boulder, CO) in 2013. Bulk DUK-CPG-001 has been resuspended in normal saline with a final concentration of 10 mg/mL, aliquoted into 0.75 mL (7.5 mg) per tube and stored at -20oC in the Investigational Chemotherapy Service pharmacy at Duke. DUK-CPG-001 will be thawed at room temperature right before use and injected intravenously right after NK cell-enriched DLI. The drug will be used within 4 hours of thawing.
  On the day of NK cell-enriched DLI, for those patients who are randomized to receive DUK-CPG-001, 0.5 mL (5 mg) aliquots of DUK-CPG-001 will be dispensed to nurse. It will be thawed at room temperature right before use and injected intravenously right after NK cell-enriched DLI.
Period: Overall Study
Arm/Group | Cohort A - NK Cell Enriched-DLI Only | Cohort A - NK-DLI + DUK-CPG-001 | Cohort B - NK Cell Enriched-DLI Only | Cohort B - NK-DLI + DUK-CPG-001
Started | 14 | 11 | 4 | 7
Completed | 7 | 5 | 0 | 2
Not Completed | 7 | 6 | 4 | 5
Not completed — Physician Decision | 4 | 4 | 3 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — still in follow-up | 2 | 2 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A - NK Cell Enriched-DLI Only | Cohort A - NK-DLI + DUK-CPG-001 | Cohort B - NK Cell Enriched-DLI Only | Cohort B - NK-DLI + DUK-CPG-001 | Total
Number analyzed (Participants) | 14 | 11 | 4 | 7 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 9 | 4 | 5 | 31
  >=65 years | 1 | 2 | 0 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 2 | 2 | 8
  Male | 11 | 10 | 2 | 5 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 11 | 10 | 2 | 7 | 30
  Unknown or Not Reported | 2 | 1 | 2 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 3 | 1 | 1 | 9
  White | 10 | 8 | 2 | 6 | 26
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 14 | 11 | 4 | 7 | 36

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Rate
Description: To evaluate the one-year progression-free survival rate in patients receiving NK cell-enriched DLI administered alone from a 7-8/8 HLA-matched related or unrelated donor or 4-6/8 HLA-matched related donor following reduced intensity or non-ablative allogeneic stem cell transplantation and to evaluate the one-year progression-free survival rate in patients receiving NK cell-enriched DLI administered with a Toll-like receptor 9 (TLR9) ligand, DUK-CPG-001, from a 7-8/8 HLA-matched related or unrelated donor or 4-6/8 HLA-matched related donor following reduced intensity or non-ablative allogeneic stem cell transplantation
Time Frame: Up to 1 year
Population: Data not collected on 13 participants.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort A - NK Cell Enriched-DLI Only | Cohort A - NK-DLI + DUK-CPG-001 | Cohort B - NK Cell Enriched-DLI Only | Cohort B - NK-DLI + DUK-CPG-001
Number analyzed (Participants) | 8 | 6 | 4 | 5
proportion of participants | 0.75 [0.31 to 0.93] | 1.00 [1.00 to 1.00] | 0.50 [0.06 to 0.84] | 0.80 [0.20 to 0.97]
Statistical Analysis 1: Comparison: Cohort A - NK Cell Enriched-DLI Only vs Cohort A - NK-DLI + DUK-CPG-001 vs Cohort B - NK Cell Enriched-DLI Only vs Cohort B - NK-DLI + DUK-CPG-001; Test type: Superiority; p = 0.40, Log Rank

2. Primary Outcome: Number of Participants With Unacceptable Toxicity
Description: Unacceptable toxicity is defined as any of the following related to the DLI procedure:
  1. Grade > III aGVHD of the gut or liver or Grade IV aGVHD of the skin lasting > 7 days;
  2. Grade 4 toxicity from the procedure in the cardiac, dermatologic, gastrointestinal, hepatic, pulmonary, renal/genitourinary, or neurologic categories that lasts > 5 days;
  3. Treatment-related death caused by the toxicities related to DLI procedure.
Time Frame: Up to 100 days
Population: Data not collected on 13 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A - NK Cell Enriched-DLI Only | Cohort A - NK-DLI + DUK-CPG-001 | Cohort B - NK Cell Enriched-DLI Only | Cohort B - NK-DLI + DUK-CPG-001
Number analyzed (Participants) | 8 | 6 | 4 | 5
Participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Recovery of Immune Cell Populations Pre and Post-Infusion
Description: To evaluate the recovery of immune cell populations pre and post infusion in patients receiving NK cell-enriched DLI administered alone or administered with TLR9 ligand, DUK-CPG-001.
Time Frame: Up to 100 days
Reporting Status: Not Posted, anticipated posting 2024-10

4. Secondary Outcome: Immune Function Pre and Post-Infusion With Antigen Specific Recovery, as Measured by Elispot Assay
Description: Pre and post infusion immune function will be reported in patients receiving NK cell-enriched DLI administered alone or administered with TLR9 ligand, DUK-CPG-001.
Time Frame: Up to 100 days
Population: Analysis of samples was not and never will be conducted, data was not collected for this Outcome Measure.
Arm/Group | Cohort A - NK Cell Enriched-DLI Only | Cohort A - NK-DLI + DUK-CPG-001 | Cohort B - NK Cell Enriched-DLI Only | Cohort B - NK-DLI + DUK-CPG-001
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Immune Function Pre and Post-Infusion With Antigen Specific Recovery, as Measured by Immunoscope Assay
Description: as for outcome 4
Time Frame: Up to 100 days
Population: Analysis of samples was not and never will be conducted, data was not collected for this Outcome Measure.
Arm/Group | Cohort A - NK Cell Enriched-DLI Only | Cohort A - NK-DLI + DUK-CPG-001 | Cohort B - NK Cell Enriched-DLI Only | Cohort B - NK-DLI + DUK-CPG-001
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Immune Function Pre and Post-Infusion With Antigen Specific Recovery, as Measured by Flow-cytometric Cytokine Assay
Description: as for outcome 4
Time Frame: Up to 100 days
Population: Analysis of samples was not and never will be conducted, data was not collected for this Outcome Measure.
Arm/Group | Cohort A - NK Cell Enriched-DLI Only | Cohort A - NK-DLI + DUK-CPG-001 | Cohort B - NK Cell Enriched-DLI Only | Cohort B - NK-DLI + DUK-CPG-001
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Immune Function Pre and Post-Infusion With Antigen Specific Recovery, as Measured by Functional NK Lysis Assay
Description: as for outcome 4
Time Frame: Up to 100 days
Population: Analysis of samples was not and never will be conducted, data was not collected for this Outcome Measure.
Arm/Group | Cohort A - NK Cell Enriched-DLI Only | Cohort A - NK-DLI + DUK-CPG-001 | Cohort B - NK Cell Enriched-DLI Only | Cohort B - NK-DLI + DUK-CPG-001
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 12 months
Arm/Group | Cohort A - NK Cell Enriched-DLI Only | Cohort A - NK-DLI + DUK-CPG-001 | Cohort B - NK Cell Enriched-DLI Only | Cohort B - NK-DLI + DUK-CPG-001
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/11 | 0/4 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/14 | 0/11 | 0/4 | 0/7
Other Adverse Events (participants affected / at risk) | 14/14 | 11/11 | 4/4 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A - NK Cell Enriched-DLI Only (N=14) | Cohort A - NK-DLI + DUK-CPG-001 (N=11) | Cohort B - NK Cell Enriched-DLI Only (N=4) | Cohort B - NK-DLI + DUK-CPG-001 (N=7)
Papilledema (Eye disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A - NK Cell Enriched-DLI Only (N=14) | Cohort A - NK-DLI + DUK-CPG-001 (N=11) | Cohort B - NK Cell Enriched-DLI Only (N=4) | Cohort B - NK-DLI + DUK-CPG-001 (N=7)
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1 | 0 | 2
Alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 2
Anemia (Blood and lymphatic system disorders) | 7 | 3 | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0
Blurred vision (Eye disorders) | 1 | 1 | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0 | 2
Creatinine increased (Investigations) | 4 | 0 | 0 | 1
Depression (Psychiatric disorders) | 3 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 1 | 0 | 0
Dry eye (Eye disorders) | 2 | 2 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 1 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Edema limbs (General disorders) | 1 | 3 | 0 | 3
Eye disorders - Other, specify (Eye disorders) | 0 | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 4 | 4 | 0 | 2
Fever (General disorders) | 0 | 1 | 0 | 1
Floaters (Eye disorders) | 0 | 2 | 0 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 5 | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 7 | 5 | 2 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 5 | 0 | 0 | 2
Hyponatremia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 2 | 0 | 0 | 0
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 1
Investigations - Other, specify (Investigations) | 1 | 2 | 0 | 2
Libido decreased (Psychiatric disorders) | 0 | 1 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 1
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 1
Neutrophil count decreased (Investigations) | 4 | 1 | 0 | 3
Obesity (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 2 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Papilledema (Eye disorders) | 1 | 0 | 0 | 0
Paresthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 2 | 0 | 2
Platelet count decreased (Investigations) | 4 | 4 | 0 | 2
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 2
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 | 0 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 3
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Retinal detachment (Eye disorders) | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 | 4 | 0 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Skin infection (Infections and infestations) | 0 | 2 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 1 | 0 | 0
Stroke (Nervous system disorders) | 0 | 1 | 0 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory infection (Infections and infestations) | 3 | 1 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 3 | 0 | 2
Urinary urgency (Renal and urinary disorders) | 1 | 2 | 0 | 0
Vascular disorders - Other, specify (Vascular disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Watering eyes (Eye disorders) | 0 | 1 | 0 | 0
Weight gain (Investigations) | 1 | 0 | 0 | 0
Weight loss (Investigations) | 1 | 2 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
White blood cell decreased (Investigations) | 5 | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-28): https://cdn.clinicaltrials.gov/large-docs/97/NCT02452697/Prot_SAP_000.pdf